CLINICAL TRIAL: NCT02739191
Title: Negative Pressure Wound Therapy for Surgical Wounds of the Foot and Ankle
Acronym: NEWTON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: J.C. Goslings (Other)
Responsible Party: Sponsor-Investigator, J.C. Goslings, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: METC 2015_280
Record Dates: First submitted 2016-04-09; First posted 2016-04-15 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Negative Pressure Wound Therapy; Vacuum Therapy; Closed Incisions
Keywords: NPWT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Prophylactic negative pressure wound therapy
  Interventions: Device: PICO, Smith & Nephew

INTERVENTIONS:
Device: PICO, Smith & Nephew — Direct application of negative pressure wound therapy following Foot and Ankle surgery

SUMMARY:
Prophylactic use of Negative Pressure Wound Therapy (NPWT) on surgical wounds following lower extremity orthopedic trauma to prevent infectious complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 and ≤ 80 years
* Orthopedic (trauma) surgery to the foot and/or ankle
* Incision >3 cm

Exclusion Criteria:

* Open fractures
* Antibiotic treatment at the time of the operation for a concomitant disease or infection
* Insufficient comprehension of the Dutch language
* Patients with immune-deficiencies
* Inability to address negative pressure wound therapy device
* Active infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04; Primary Completion 2017-03 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Number patients with postoperative wound infections (POWI) as classified bij the Centers for Disease Control and prevention (CDC)-criteria. | 30 days
  The number of POWI's within 30 days of surgery will be recorded. These will be classified in superficial and deep POWI's using the criteria as proposed by the CDC.

SECONDARY OUTCOMES:
The American Orthopaedic Foot and Ankle Score (AOFAS) will be measured at six months | 6 months
  To asses functional outcome of the participants the AOFAS questionnaire will be used
EuroQol five dimensions questionnaire (EQ-5D)will be measured at six months | 6 months
  To asses the quality of life of the participants the EQ-5D questionnaire will be used

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands